CLINICAL TRIAL: NCT05989815
Title: Effect of Whole-body Photobiomodulation on Muscular Performance Enhancement.
Acronym: WBPME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Italo Amaral de Oliveira, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 62842522.2.0000.5504
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Sports Performance; Injury Prevention; Muscle Damage; Musculoskeletal Pain
Keywords: phototherapy; laser therapy; muscle fatigue; muscle damage
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PBMT post muscle damage protocol (PBMT-post) (Experimental): Group submitted to pre-exercise Sham (placebo) photobiomodulation therapy (PBMT), and post-exercise active PBMT.
  PBMT will be administered using a whole-body irradiation system (Joovv Elite System, Joovv Inc.), consisting of 6 panels with 76 red LEDs (660 ± 10 nm) and 74 infrared LEDs (850 ± 10 nm), totaling 900 LEDs covering an area of 12,193 cm². Athletes will stand 20 cm in front of the device, wearing only swim shorts to expose their thigh muscles and other body areas to the light. The total irradiation time will be 20 minutes, with 10 minutes (600 seconds) of irradiation for the anterior region and another 10 minutes (600 seconds) for the posterior region. The active PBMT dose applied in each region (anterior or posterior) will be 48.97 J/cm², with an irradiance of 81.62 mW/cm².
  Interventions: Other: Muscle damage protocol training; Device: Photobiomodulation therapy (PBMT)
- PBMT pre (PBMT-pre) (Experimental): Group submitted to pre-exercise active photobiomodulation therapy (PBMT), and post-exercise Sham (placebo) PBMT.
  PBMT will be administered using a whole-body irradiation system (Joovv Elite System, Joovv Inc.), consisting of 6 panels with 76 red LEDs (660 ± 10 nm) and 74 infrared LEDs (850 ± 10 nm), totaling 900 LEDs covering an area of 12,193 cm². Athletes will stand 20 cm in front of the device, wearing only swim shorts to expose their thigh muscles and other body areas to the light. The total irradiation time will be 20 minutes, with 10 minutes (600 seconds) of irradiation for the anterior region and another 10 minutes (600 seconds) for the posterior region. The active PBMT dose applied in each region (anterior or posterior) will be 48.97 J/cm², with an irradiance of 81.62 mW/cm².
  Interventions: Other: Muscle damage protocol training; Device: Photobiomodulation therapy (PBMT)
- PBMT placebo (PBMT-sham) (Sham Comparator): Group submitted to pre-exercise and post-exercise photobiomodulation therapy (PBMT) Sham (placebo).
  PBMT will be administered using a whole-body irradiation system (Joovv Elite System, Joovv Inc.), consisting of 6 panels with 76 red LEDs (660 ± 10 nm) and 74 infrared LEDs (850 ± 10 nm), totaling 900 LEDs covering an area of 12,193 cm². Athletes will stand 20 cm in front of the device, wearing only swim shorts to expose their thigh muscles and other body areas to the light. The total irradiation time will be 20 minutes, with 10 minutes (600 seconds) of irradiation for the anterior region and another 10 minutes (600 seconds) for the posterior region. The Sham PBMT dose applied in each region (anterior or posterior) will be 0 J/cm², with an irradiance of 0 mW/cm².
  Interventions: Other: Muscle damage protocol training; Device: Photobiomodulation therapy (PBMT)

INTERVENTIONS:
Other: Muscle damage protocol training — The adopted protocol of muscle damage will follow the recommendations from American College of Sports Medicine (ACSM) in 2009 for trained individuals. It consists of 8-12 repetitions above 70% of 1 Repetition Maximum (1RM) with 1 minute of rest between sets and 2 minutes between exercises. The protocol will be composed as follows: 3 sets of 10 repetitions for each exercise, with an emphasis on producing microlesions in the muscle tissue (muscle damage protocol).
Device: Photobiomodulation therapy (PBMT) — PBMT will be administered using a whole-body irradiation system (Joovv Elite System, Joovv Inc.), consisting of 6 panels with 76 red LEDs (660 ± 10 nm) and 74 infrared LEDs (850 ± 10 nm), totaling 900 LEDs covering an area of 12,193 cm². Athletes will stand 20 cm in front of the device, wearing only swim shorts to expose their thigh muscles and other body areas to the light. The total irradiation time will be 20 minutes, with 10 minutes (600 seconds) of irradiation for the anterior region and another 10 minutes (600 seconds) for the posterior region. The active PBMT dose applied in each region (anterior or posterior) will be 48.97 J/cm², with an irradiance of 81.62 milliwatt (mW)/cm². The PBMT Sham dose applied in each region (anterior or posterior) will be 0 J/cm², with an irradiance of 0 mW/cm².

SUMMARY:
Introduction: Photobiomodulation therapy (PBMT) is based on the emission of light ranging from red to near-infrared spectra by different devices based on diode lasers or light-emitting diodes. These devices emitting different wavelengths can increase mitochondrial activity and energy synthesis (ATP - adenosine triphosphate) that in turn can help to prevent muscle damage, decrease muscle fatigue and enhance muscle performance. Thus, PBMT can be a promising therapeutic resource in the sports field. Objectives: The aim of this study is to verify the effect of PBMT on the muscle performance and prevention of muscle damage and delayed onset muscle soreness (DOMS) in professional soccer players submitted to a muscle damage protocol. Methodology: The present study is a randomized sham-controlled clinical trial following the CONSORT guidelines.

DETAILED DESCRIPTION:
Participants will be allocated into 3 balanced randomized groups, as follows: 1) PBMT post muscle damage protocol (PBMT-post); 2) PBMT pre (PBMT-pre) and 3) PBMT placebo (PBMT-sham). All groups will be submitted to a) anamnesis; b) measurement of blood levels of creatine phosphokinase (CK); c) delayed onset muscle soreness (DOMS); d) muscle performance tests (Squat Jump test (SJ) and Counter Movement Jump (CMJ)); e) dynamometry of the knee extensor muscles. Whole body PBMT will be applied according to the groups, during 10 min (sham or effective), with an effective dose of 48.97 J/cm2 and irradiance of 81.62 mW/cm2. Muscle damage protocol will consist of 8 exercises for lower limb muscles, with 3 sets of 10 repetitions each, 1 minute of rest between sets, and 2 minutes of rest between exercises. Next, participants will be evaluated for levels of CK, DOMS and muscle performance (SJ, CMJ, dynamometry) at 24, 48 and 72 hours after muscle damage protocol. Data will be analyzed and compared between groups with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged between 18 and 35 years, professional soccer players who engage in training at least 5 times a week, will be selected.

Data collection will be conducted at the Desportivo Brasil Football Club, located in Porto Feliz, São Paulo. The sample will consist of team members, with a total of 30 athletes established to compose the sample. All data collection will take place in the same location.

Exclusion Criteria:

* Individuals with any impediment to physical activity or those presenting dysfunctions that may impair the neuromuscular system will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Ferraresi, Phd, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Desportivo Brasil Football Club, Porto Feliz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zagatto AM, Dutra YM, Lira FS, Antunes BM, Faustini JB, Malta ES, Lopes VHF, de Poli RAB, Brisola GMP, Dos Santos GV, Rodrigues FM, Ferraresi C. Full Body Photobiomodulation Therapy to Induce Faster Muscle Recovery in Water Polo Athletes: Preliminary Results. Photobiomodul Photomed Laser Surg. 2020 Dec;38(12):766-772. doi: 10.1089/photob.2020.4803. PMID 33332232
- [Background] Thong ISK, Tan G, Lee TYC, Jensen MP. A Comparison of Pain Beliefs and Coping Strategies and Their Association with Chronic Pain Adjustment Between Singapore and United States. Pain Med. 2017 Sep 1;18(9):1668-1678. doi: 10.1093/pm/pnw237. PMID 27694147
- [Background] Lesnak J, Anderson D, Farmer B, Katsavelis D, Grindstaff TL. VALIDITY OF HAND-HELD DYNAMOMETRY IN MEASURING QUADRICEPS STRENGTH AND RATE OF TORQUE DEVELOPMENT. Int J Sports Phys Ther. 2019 Apr;14(2):180-187. PMID 30997270
- [Background] Higashi RH, Toma RL, Tucci HT, Pedroni CR, Ferreira PD, Baldini G, Aveiro MC, Borghi-Silva A, de Oliveira AS, Renno AC. Effects of low-level laser therapy on biceps braquialis muscle fatigue in young women. Photomed Laser Surg. 2013 Dec;31(12):586-94. doi: 10.1089/pho.2012.3388. PMID 24320801
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Psychometric properties of the portuguese version of the Pain Self-Efficacy Questionnaire. Acta Reumatol Port. 2011 Jul-Sep;36(3):260-7. PMID 22113601
- [Background] Enwemeka CS. Light is light. Photomed Laser Surg. 2005 Apr;23(2):159-60. doi: 10.1089/pho.2005.23.159. No abstract available. PMID 15910178
- [Background] Denadai AS, de Carvalho Pde T, dos Reis FA, Belchior AC, Pereira DM, Dourado DM, Silva IS, de Oliveira LV. Morphometric and histological analysis of low-power laser influence on bone morphogenetic protein in bone defects repair. Lasers Med Sci. 2009 Sep;24(5):689-95. doi: 10.1007/s10103-008-0595-6. Epub 2008 Sep 12. PMID 18787760
- [Background] Dornelles MP, Fritsch CG, Sonda FC, Johnson DS, Leal-Junior ECP, Vaz MA, Baroni BM. Photobiomodulation therapy as a tool to prevent hamstring strain injuries by reducing soccer-induced fatigue on hamstring muscles. Lasers Med Sci. 2019 Aug;34(6):1177-1184. doi: 10.1007/s10103-018-02709-w. Epub 2019 Jan 3. PMID 30607719
- [Background] Cressoni MD, Dib Giusti HH, Casarotto RA, Anaruma CA. The effects of a 785-nm AlGaInP laser on the regeneration of rat anterior tibialis muscle after surgically-induced injury. Photomed Laser Surg. 2008 Oct;26(5):461-6. doi: 10.1089/pho.2007.2150. PMID 18800950
- [Background] Azuma RHE, Merlo JK, Jacinto JL, Borim JM, da Silva RA, Pacagnelli FL, Nunes JP, Ribeiro AS, Aguiar AF. Photobiomodulation Therapy at 808 nm Does Not Improve Biceps Brachii Performance to Exhaustion and Delayed-Onset Muscle Soreness in Young Adult Women: A Randomized, Controlled, Crossover Trial. Front Physiol. 2021 Jun 10;12:664582. doi: 10.3389/fphys.2021.664582. eCollection 2021. PMID 34177615
- [Background] Julio CE, Antonialli FC, Nascimento TMD, Sa KA, Barton GJ, Lucareli PRG. The Movement Deviation Profile Can Differentiate Faller and Non-Faller Older Adults. J Gerontol A Biol Sci Med Sci. 2023 Aug 27;78(9):1651-1658. doi: 10.1093/gerona/glad141. PMID 37279546
- [Background] Anders JJ, Arany PR, Baxter GD, Lanzafame RJ. Light-Emitting Diode Therapy and Low-Level Light Therapy Are Photobiomodulation Therapy. Photobiomodul Photomed Laser Surg. 2019 Feb;37(2):63-65. doi: 10.1089/photob.2018.4600. Epub 2019 Jan 24. No abstract available. PMID 31050924
- [Background] Qureshi MA, Mcisaac L, Schlyer D, Hupf HB, Al-Watban FA, Lewall D. Production of 123I as iodide by distillation. Int J Nucl Med Biol. 1985;12(1):57-8. doi: 10.1016/0047-0740(85)90014-2. No abstract available. PMID 4008167
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with injuries that prevented them from practicing sports were excluded.
Groups:
- PBMT Post Muscle Damage Protocol (PBMT-post): Group submitted to pre-exercise Sham (placebo) photobiomodulation therapy (PBMT), and post-exercise active PBMT.
- PBMT Pre (PBMT-pre): Group submitted to pre-exercise active photobiomodulation therapy (PBMT), and post-exercise Sham (placebo) PBMT.
- PBMT Placebo (PBMT-sham): Group submitted to pre-exercise and post-exercise photobiomodulation therapy (PBMT) Sham (placebo).
Period: Overall Study
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were professional male soccer players (18-35 years) from the same training team.
  Baseline demographic and anthropometric data were collected prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 20 (1) | 20 (1) | 20 (1) | 20 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Blood Levels of Creatine Phosphokinase (CK)
Description: Mean serum creatine phosphokinase (CK) concentration (U/L), calculated as the average of four time points: Baseline, 24h, 48h, and 72h post-exercise. Higher values indicate greater muscle damage.
Time Frame: Average of Baseline, 24h, 48h, and 72h
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Number analyzed (Participants) | 10 | 10 | 10
U/L | 287.8 (199.09) | 249.2 (112.28) | 289.2 (209.94)

2. Secondary Outcome: Squat Jump (SJ) Height
Description: Vertical jump height (cm) measured by the Squat Jump (SJ) test. Mean of four time points: Baseline, 24h, 48h, and 72h after the protocol. Higher values indicate better performance.
Time Frame: Average of Baseline, 24h, 48h, 72h
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Number analyzed (Participants) | 10 | 10 | 10
cm | 37.38 (5.22) | 38.91 (5.45) | 38.56 (4.09)

3. Secondary Outcome: Muscle Performance Tests - Dynamometry
Description: Peak isometric force (kgf) of knee extensors, measured with handheld dynamometry.
  Mean of Baseline, 24h, 48h, and 72h after exercise. Higher values indicate better performance.
Time Frame: Average of Baseline, 24h, 48h, and 72h
Measure: Mean (Standard Deviation); unit: kgf (kilogram-force)
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Number analyzed (Participants) | 10 | 10 | 10
kgf (kilogram-force) | 59.19 (8.34) | 53.45 (8.63) | 55.58 (10.45)

4. Secondary Outcome: Delayed Onset Muscle Soreness (DOMS)
Description: DOMS intensity assessed using a Numeric Rating Scale (NRS; 0-10), where 0 = no soreness and 10 = worst possible soreness during knee extension. Higher scores indicate greater soreness. Mean of Baseline, 24h, 48h, and 72h post-protocol.
Time Frame: Average of Baseline, 24h, 48h, and 72h
Measure: Mean (Standard Deviation); unit: points on NRS (0-10)
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Number analyzed (Participants) | 10 | 10 | 10
points on NRS (0-10) | 3.00 (2.00) | 3.80 (2.74) | 5.70 (2.05)

5. Secondary Outcome: Countermovement Jump (CMJ) Height
Description: Vertical jump height (cm) measured by the Countermovement Jump (CMJ) test. Mean of four time points: Baseline, 24h, 48h, and 72h after the protocol. Higher values indicate better performance.
Time Frame: Average of Baseline, 24h, 48h, 72h
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
Number analyzed (Participants) | 10 | 10 | 10
cm | 39.36 (4.27) | 41.56 (6.73) | 40.55 (4.28)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 4 consecutive days, from baseline through 72 hours post-protocol.
Description: Adverse events were monitored and recorded using standard definitions aligned with ClinicalTrials.gov. No deviation from the standard definitions of adverse event or serious adverse event occurred. Participants were systematically questioned and observed during all evaluation sessions across the 4-day study period.
Arm/Group | PBMT Post Muscle Damage Protocol (PBMT-post) | PBMT Pre (PBMT-pre) | PBMT Placebo (PBMT-sham)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT05989815/Prot_SAP_002.pdf